CLINICAL TRIAL: NCT03557489
Title: Effectiveness of Sacral Foam Pad in Preventing Pressure Injury in Surgical Patients With Supine Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, MAH CHUN, Deputy Director of Nursing Department, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107HCP-08
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients use gel pad(in usual) in addition to(Mepilex Border Sacrum)foam pad during surgery.
  Interventions: Device: Mepilex Border Sacrum
- Control group (No Intervention): patients use gel pad(in usual) during surgery.

INTERVENTIONS:
Device: Mepilex Border Sacrum — Patients use gel pad(in usual) in addition to use Mepilex Border Sacrum foam pad during surgery.
  Arms: Experimental group

SUMMARY:
In surgical patients, prevention of pressure injury is a challenge because of the high risk for multiple comorbid conditions, hemodynamic instability, and long duration of immobility.

The objectives of our study is to compare the difference in incidence rates of sacral pressure injury in surgical patients with supine position more than 3 hours between those treated with usual preventive care and a sacral foam pad versus a control group receiving usual care.

DETAILED DESCRIPTION:
The incidence of pressure injury in surgical patients about 12% to 45%, though these patients were treated with "gel pad" as routine. Based on the nutritional status of patients, long-term surgery, surgical posture, and anesthesia-induced hypotension, pressure injury still occurred. Sacral foam pad (Mepilex(®) Border Sacrum) is an unique 5-layer design, was designed to protect sacral pressure injury. In this study, we enrolled surgical patients who need to supine over ≧ 3 hours to evalute the effectiveness of sacral foam pad in preventing sacral pressure injury. The patients will randomized to control and intervention groups, both groups recruited 105 patients. In control group, patients use gel pad during surgery; whereas patients use gel pad in addition to sacrum foam pad (Mepilex(®) Border Sacrum) in intervention group. After surgery, the occurrence and severity of sacral pressure injury was evaluated. The results of this study can provide evidence to improve the awareness of operating room medical staff on surgical pressure injury, and find out the risk factors in avoiding of pressure injury, and offer an effective strategy to enhance the quality of surgery throughout the perioperative care.

ELIGIBILITY:
Inclusion Criteria:

1.20-99 years old surgical patients who need to supine position over ≧ 3 hours 2.Patients have no any skin lesion.

Exclusion Criteria:

1. under 20 years
2. Patients have any skin lesion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-06-16 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Sacral pressure injury | After 1 hour surgery
  After surgery check patient's sacral skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Chun Mah, MS, Principal Investigator — Deputy Director of Nursing Department in Shuang Ho Hospital

IPD SHARING:
Plan to Share IPD: Undecided